CLINICAL TRIAL: NCT00117585
Title: Orthostatic Hypotension in Rehabilitation Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E3616-R
Record Dates: First submitted 2005-06-30; First posted 2005-07-07 (Estimated); Results first posted 2014-07-04 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-03

CONDITIONS: Hypotension, Orthostatic
Keywords: Aging; Blood pressure; Hypotension; Orthostatic; Rehabilitation
MeSH Terms: conditions — Hypotension, Orthostatic; Hypotension | interventions — fludrocortisone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Phase 1 (Other): Stepped intervention consisting of treatment phase 1, 2 and 3. Subjects whose orthostatic hypotension is resolved after treatment phase 1 will not receive new treatments (phase 2 and 3)
  Interventions: Other: Treatment Phase 1; Drug: Treatment Phase 2; Other: Treatment Phase 3

INTERVENTIONS:
Other: Treatment Phase 1 — * Patient Education
  * Physical Therapy Exercises
  * Increased Salt Intake
  * Elevation of head of bed with 2-4 inch wedge
  * Medication Review by MD, Pharma
Drug: Treatment Phase 2 — Subjects receive Treatment Phase 2 if they are still orthostatic after receiving Treatment Phase 1.
  * Fludrocortisone
  * Salt tablet
  Other Names: Florinef
Other: Treatment Phase 3 — Subjects still experiencing orthostatic hypotension after receiving Treatment Phases 1 and 2 move on to Treatment Phase 3. Individualized treatment is based on subspecialty or orthostatic hypotension consultation at the medical center. Subjects are followed for the duration of their hospital stay, on average 4 weeks.

SUMMARY:
The purpose of this study is to determine the prevalence and clinical course of orthostatic hypotension (OH) on a rehabilitation and nursing home unit during their inpatient stay and to initiate a standardized, interdisciplinary treatment plan for patients with OH and determine the effect of treatment on the clinical course of OH during their inpatient stay.

DETAILED DESCRIPTION:
This study is a prospective, quasi-experiment conducted in two consecutive phases. During the observation phase, eligible patients are identified and followed through their usual course of care in the nursing home/rehabilitation unit. During the intervention phase, patients enrolled who have OH will receive the intervention. Patients will be enrolled over two research phases and the investigators expect to evaluate 459 subjects. This research program will occur over a three-year period.

Methods:

During Phase I, baseline prevalence and natural history of OH will be determined by: enrolling consecutive appropriate subjects (able to stand, not end of life care) from a rehabilitation and nursing home unit and measuring OH 3 times weekly over their inpatient stay. In addition, chart review of diagnoses, medications, functional status, nutrition, and adverse events will be evaluated and correlated with clinical status. During Phase II, the investigators will implement a standardized, interdisciplinary (MD/RN/PT/Dietician) treatment plan for patients with OH. This will include chart review of diagnoses, medications, functional status, nutrition, adverse events, and correlation with clinical status. The goals of the interventions are to identify and treat the underlying causes of OH in rehabilitation patients. Based upon the comprehensive assessment, intervention participants will receive a standardized, interdisciplinary treatment regime.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to Vancouver VA Nursing Home or Rehabilitation ward

Exclusion Criteria:

* Unable to stand upon admission
* Hospice admission
* Respite admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 341 (Actual)
Dates: Start 2005-11; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- VA Portland Health Care System, Portland, OR, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 341 subjects were recruited. These subjects were recruited from all admits to the rehabilitation unit.
Pre-assignment Details: Exclusion criteria included subjects who: couldn't stand, were admitted for respite, and were anticipated to only be on station for less than 7 days.
Groups:
- Arm 1: Stepped intervention consisting of three treatment phases
  Treatment 1 :
  Patient Education Physical Therapy Exercises Increased Salt Intake Elevation of head of bed with 2-4 inch wedge Medication Review by MD, Pharmacist
  Treatment 2 : Fludrocortisone Salt tablets
  Treatment 3 : Individualized treatment based on subspecialty or orthostatic hypotension consultation at the medical center
Period: Overall Study
Arm/Group | Arm 1
Started | 341
Completed | 341
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1
Number analyzed (Participants) | 341
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 341
Age, Continuous [Mean (Standard Deviation); unit: years] | 75 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 300
Region of Enrollment [Number; unit: participants]
  United States | 341

OUTCOME MEASURES:

1. Primary Outcome: Orthostatic Hypotension at Discharge
Description: Participants are assessed for orthostatic hypotension up to one time per day. The outcome measure is the last three days prior to discharge that blood pressures were assessed for orthostatic hypotension.
Time Frame: Last three blood pressures prior to discharge
Measure: Number; unit: participants
Arm/Group | Arm 1
Number analyzed (Participants) | 341
participants | 96

ADVERSE EVENTS:
Arm/Group | Arm 1
Serious Adverse Events (participants affected / at risk) | 6/341
Other Adverse Events (participants affected / at risk) | 0/341
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=341)
Death (General disorders) | 6 — Death is not an unexpected SAE in this nursing home population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes